CLINICAL TRIAL: NCT00598624
Title: Clinical Phase II Trial to Evaluate the Safety and Efficacy of Treosulfan Based Conditioning Prior to Allogeneic Haematopoietic Stem Cell Transplantation in Patients With Haematological Malignancies
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of Treosulfan Based Conditioning Prior to Allogeneic Haematopoietic Stem Cell Transplantation (HSCT)
Acronym: AlloTreo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Fabio Ciceri, MD, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-005182-11
Record Dates: First submitted 2008-01-10; First posted 2008-01-22 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Leukemia; Chronic Myeloid Leukemia; Myelodysplastic Syndrome; Diffuse Large Cell Lymphoma; Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Multiple Myeloma
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Treosulfan IV

INTERVENTIONS:
Drug: Treosulfan IV — Treosulfan i.v.: 14 g/m²/d from day -6 to day -4

SUMMARY:
This is a multicentric, non-randomized, non-controlled open-label phase II trial to evaluate the safety and efficacy of treosulfan in a combination regimen with fludarabine as conditioning therapy prior to allogeneic stem cell transplantation (SCT) in patients with haematological malignancies.

The aim is to demonstrate a clinical benefit compared with historical data on intravenous busulfan (BusulfexTM, BusilvexTM), the only drug so far registered in the indication conditioning before allogeneic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with haematological malignancies, according to WHO classification, such as:

   * acute myeloid leukaemia -AML- in CR1 except "low-risk cases" defined by t(15;17), t(8;21), inv 16 or normal cytogenetics at diagnosis with FLT3-ITD negative and NPM-1 positive, with no high risk clinical criteria
   * any AML beyond CR1
   * acute lymphoblast leukaemia -ALL- in CR1 only if at "high risk" defined by cytogenetics as t(9;22), t(4;11) or for persistence of minimal residual disease (MRD)
   * any ALL beyond CR1
   * chronic myeloid leukaemia -CML- in chronic phase (CP) or accelerated phase (AP) intolerant/not responsive to TK-inhibitors
   * myeloproliferative disorders -MPD-
   * myelodysplastic syndrome -MDS- with intermediate or high risk International Prognostic Scoring System (IPSS)
   * diffuse large cell lymphoma -DLCL- with a chemosensitive relapse or beyond CR1
   * lymphoblastic and Burkitt lymphoma with a chemosensitive relapse or beyond CR1
   * mantle cell lymphoma -MCL- with a chemosensitive relapse or beyond CR1
   * follicular lymphoma -FCL- with a chemosensitive relapse or beyond CR2
   * Hodgkin lymphoma -HD- with a chemosensitive relapse or beyond CR1
   * chronic lymphocytic leukaemia -CLL- at "poor risk" in CR1 or with a chemosensitive relapse
   * CLL relapsing after high dose chemotherapy
   * T-cell non Hodgkin lymphoma -T-NHL- in CR1 or beyond
   * multiple myeloma -MM- at high risk for cytogenetics or ISS stage 3 in CR1 following high dose chemotherapy
   * MM at any relapse/progression except refractory disease
2. Availability of an HLA-identical sibling donor (MRD) or HLA-identical unrelated donor (MUD)

   * HLA-identity defined by the following markers: A, B, DRB1, DQB1 or a single or double Cord Blood unit (CB) with at least a 4 out of 6 HLA-matching by the following markers: A, B and DRB.

   A) identity between the 2 CB units and the recipient;

   B) Two identical CB units with one or two mismatches with the recipient;

   C) Two CB units with one mismatch between them and two mismatches with the recipient. We will prefer mismatches either for class I or for class II antigens; we will avoid mismatches concerning both classes I and II together.
3. Target graft size (unmanipulated, preferably not cryopreserved)

   * bone marrow: 2 to 10 x 106 CD34+ cells/kg BW recipient or > 2 x 108 nucleated cells/kg BW recipient or
   * peripheral blood: 4 to 10 x 106 CD34+ cells/kg BW recipient
4. Age > 18 and < 70 years
5. Karnofsky Index > 80 %
6. Adequate contraception in female patients of child-bearing potential
7. Written informed consent

Exclusion Criteria:

1. Secondary malignancies
2. Previous allogeneic transplantation
3. Hematopoietic cell transplantation-specific comorbidity index > 4 (HCT-CI Sorror et al, Appendix M)
4. Known and manifested malignant involvement of the CNS
5. Active infectious disease
6. HIV- positivity or active hepatitis infection
7. Impaired liver function (Bilirubin > upper normal limit; Transaminases > 3.0 x upper normal limit)
8. Impaired renal function (Creatinine-clearance < 60 ml/min; Serum Creatinine > 1.5 x upper normal limit).
9. Pleural effusion or ascites > 1.0 L
10. Pregnancy or lactation
11. Known hypersensitivity to treosulfan and/or fludarabine
12. Participation in another experimental drug trial within 4 weeks before day -6
13. Non-co-operative behaviour or non-compliance
14. Psychiatric diseases or conditions that might impair the ability to give informed consent

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Evaluation of engraftment | 28 days
Safety: Evaluation of the incidence of CTC grade 3 and 4 adverse events | between day -6 and day +28

SECONDARY OUTCOMES:
Efficacy: Evaluation of disease free survival (DFS) | 1 year
Efficacy: Evaluation of overall survival (OS) | 1 year
Efficacy: Evaluation of relapse incidence (RI) | 1 year
Efficacy: Documentation of donor chimerism | on day +28, +56 and +100
Safety: Evaluation of incidence of non-relapse mortality (NRM) | on day +28 and day +100
Safety: cumulative incidence of NRM | 1 year
Safety: Evaluation of cumulative incidence and severity of acute and chronic graft vs. host disease (GvHD) | 1 year
Safety: EBV reactivation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Fabio FC Ciceri, MD, Study Director
Locations (12):
- Italy (12):
  - Ematologia, Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - IRCCS San Raffaele; Unità Operativa di Ematologia, Milan, MI
  - Dipartimento Biotecnologie Cellulari ed Ematologia; Azienda Policlinico Umberto I, Roma, Roma
  - USC Ematologia, Ospedali Riuniti, Bergamo
  - Ospedale centrale di Bolzano - Reparto di Ematologia, Bolzano
  - PO "R.Binaghi" - CTMO, Cagliari
  - AO "Santa Croce" e Carle - Reparto di Ematologia, Cuneo
  - Istituto Europeo di Oncologia - Divisione di Ematologia, Milan
  - Ospedale Civile - UTI ematologia per il trapianto emopoietico, Pescara
  - Arcispedale Santa Maria Nuova - SC di Ematologia, Reggio Emilia
  - AO San Camillo Forlanini - UOC ematologia e trapianto, Roma
  - AOU Santa Maria della Misericordia - Clinica Ematologica, Udine

REFERENCES:
- [Derived] Lazzari L, Ruggeri A, Lupo Stanghellini MT, Mastaglio S, Messina C, Giglio F, Lorusso A, Perini T, Piemontese S, Marcatti M, Lorentino F, Xue E, Clerici D, Corti C, Bernardi M, Assanelli A, Greco R, Ciceri F, Peccatori J. Treosulfan-Based Conditioning Regimen Prior to Allogeneic Stem Cell Transplantation: Long-Term Results From a Phase 2 Clinical Trial. Front Oncol. 2021 Sep 10;11:731478. doi: 10.3389/fonc.2021.731478. eCollection 2021. PMID 34568066